CLINICAL TRIAL: NCT03936673
Title: The Effect of Percutaneous Nephrostomy Application on Obstructed Kidneys With Relative Function of 10% or Less In Technetium-99m Dimercaptosuccinic Acid (DMSA) Scintigraphy
Brief Title: Effect of Nephrostomy on Relative Function of Obstructed Kidney
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Abdullah Demirtas, Md, Assoc Prof, TC Erciyes University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014/349
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Obstructive Uropathy
Keywords: obstructive uropathy; relative renal function; DMSA
MeSH Terms: interventions — Nephrostomy, Percutaneous

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with unilateral obstructed kidney with RRF 10% or less underwent application of percutaneous nephrostomy tube on affected side.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- atrophic kidney (Experimental): Patients diagnosed with unilateral obstructed kidney with RRF 10% or less underwent application of percutaneous nephrostomy tube on affected side.
  Interventions: Procedure: Percutaneous nephrostomy

INTERVENTIONS:
Procedure: Percutaneous nephrostomy

SUMMARY:
Urinary tract obstruction is a serious health problem due to kidney damage. Relative renal function has an important role in the treatment of obstructed kidneys. Nephrectomy can be recommended when the relative renal function is 10% or less in radionuclide examinations. Recently, however, nephron sparing approaches have come to the fore. This indicated the need to evaluate the possibility of recovering the function of the kidney before nephrectomy. The aim of this study is to compare relative functions of obstructed kidneys in technetium 99m dimercaptosuccinic acid scintigraphy (DMSA) before and 2 weeks after nephrostomy tube.

DETAILED DESCRIPTION:
Obstructive uropathy is one of the most important causes of acute renal injury and end-stage renal failure. obstruction of urine flow increases the intratubular pressure. This pressure increase causes decrease in renal blood flow and starts the inflammatory process. In the first few hours after total ureter obstruction, due to the increase in intratubular pressure glomerular filtration ceases and tubular transport is markedly decreased. Long lasting obstruction results in renal fibrosis and end stage renal damage. Basically obstructive uropathy leading to irreversible renal damage and loss of renal function is the main indication for simple nephrectomy. Serious renal parenchymal damage is defined as non-functioning kidney having relative renal function (RRF) 10% or less in the literature. But recently in some studies it was suggested that by applying the nephrostomy catheter, ability of kidney to regain function can be evaluated before nephrectomy. So, possibility of gaining function should be kept in mind. In this study effect of percutaneous nephrostomy tube on serum creatinine, blood urea nitrogen (BUN) and RRF in obstructed kidney with RRF 10% or less. Before and 2 weeks after percutaneous nephrostomy, serum creatinine, ure and RRF in DMSA was recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral obstructed kidney with RRF 10% or less
* Unilateral obstructed kidney with grade 2 or more hydroureteronephrosis
* Defined etiology for unilateral obstructed kidney
* estimated glomerular filtration rate (GFR) ≥ 30ml/min
* Approving the nephrostomy procedure

Exclusion Criteria:

* Unilateral obstructed kidney with RRF above 10%
* Estimated GFR <30 ml/min
* diagnosis of bilateral obstructed kidneys
* not approving nephrostomy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
serum creatinine level 2 weeks after nephrostomy | 2 weeks after nephrostomy
  serum creatinine level 2 weeks after nephrostomy
Serum BUN level 2 weeks after nephrostomy | 2 weeks after nephrostomy
  Serum BUN level 2 weeks after nephrostomy
RRF in DMSA 2 weeks after nephrostomy | 2 weeks after nephrostomy
  RRF in DMSA 2 weeks after nephrostomy

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah T Demirtas, Assoc Prof, Principal Investigator — Erciyes University Faculty of Medicine
Locations (1):
- Department of Urology, Ercieys University, Faculty Of Medicine,, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thorup J, Jokela R, Cortes D, Nielsen OH. The results of 15 years of consistent strategy in treating antenatally suspected pelvi-ureteric junction obstruction. BJU Int. 2003 Jun;91(9):850-2. doi: 10.1046/j.1464-410x.2003.04228.x. PMID 12780846
- [Background] Gupta DK, Chandrasekharam VV, Srinivas M, Bajpai M. Percutaneous nephrostomy in children with ureteropelvic junction obstruction and poor renal function. Urology. 2001 Mar;57(3):547-50. doi: 10.1016/s0090-4295(00)01046-3. PMID 11248637
- [Background] Ismail A, Elkholy A, Zaghmout O, Alkadhi A, Elnaggar O, Khairat A, Elhassanat H, Mosleh A, Hamad B, Elzomer J, Elkaabi A. Postnatal management of antenatally diagnosed ureteropelvic junction obstruction. J Pediatr Urol. 2006 Jun;2(3):163-8. doi: 10.1016/j.jpurol.2005.07.005. Epub 2005 Aug 26. PMID 18947602
- [Background] Morduchowicz G, Winkler J, Zabludowski JR, Boner G. Effects of residual renal function in haemodialysis patients. Int Urol Nephrol. 1994;26(1):125-31. doi: 10.1007/BF02768252. PMID 8026917
- [Background] Wang AY, Wang M, Woo J, Law MC, Chow KM, Li PK, Lui SF, Sanderson JE. A novel association between residual renal function and left ventricular hypertrophy in peritoneal dialysis patients. Kidney Int. 2002 Aug;62(2):639-47. doi: 10.1046/j.1523-1755.2002.00471.x. PMID 12110029
- [Background] Bargman JM, Thorpe KE, Churchill DN. Relative contribution of residual renal function and peritoneal clearance to adequacy of dialysis: a reanalysis of the CANUSA study. J Am Soc Nephrol. 2001 Oct;12(10):2158-2162. doi: 10.1681/ASN.V12102158. PMID 11562415
- [Result] Zhang S, Zhang Q, Ji C, Zhao X, Liu G, Zhang S, Li X, Lian H, Zhang G, Guo H. Improved split renal function after percutaneous nephrostomy in young adults with severe hydronephrosis due to ureteropelvic junction obstruction. J Urol. 2015 Jan;193(1):191-5. doi: 10.1016/j.juro.2014.07.005. Epub 2014 Jul 9. PMID 25014578
- [Result] Aziz MA, Hossain AZ, Banu T, Karim MS, Islam N, Sultana H, Alam MI, Hanif A, Khan AR. In hydronephrosis less than 10 % kidney function is not an indication for nephrectomy in children. Eur J Pediatr Surg. 2002 Oct;12(5):304-7. doi: 10.1055/s-2002-35956. PMID 12469255